CLINICAL TRIAL: NCT03533309
Title: Accuracy of Computer Guided Versus Conventional Ridge Splitting of Horizontal Deficient in Maxillary Anterior Alveolar Ridge (Randomized Clinical Trial)
Brief Title: Accuracy of Computer Guided Versus Conventional Ridge Splitting of Horizontal Deficient in Maxillary Anterior Alveolar Ridge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, abdalrahman Aburas, Doctor, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 152018
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Ridge Deficency
Keywords: horizontal defect, Anterior maxillary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer guided (Experimental): Group (A): comprised 6 patient undergoing surgical alveolar ridge splitting using computer guided surgical cutting stent.
  .
  Interventions: Procedure: Computer guided surgical cutting guide
- conventional (Active Comparator): Group (B) comprised 6 patient undergoing surgical alveolar ridge splitting using conventional technique
  Interventions: Procedure: Conventional alveolar ridge splitting

INTERVENTIONS:
Procedure: Computer guided surgical cutting guide — comprised 6 patient undergoing surgical alveolar ridge splitting using computer guided surgical cutting stent
  Arms: computer guided
Procedure: Conventional alveolar ridge splitting — comprised 6 patient undergoing surgical alveolar ridge splitting using conventional technique.
  Arms: conventional

SUMMARY:
In patient with horizontal deficiency in alveolar ridge of the anterior maxilla, Dose computer Guided stent enhance the accuracy and clinical outcome vs conventional ridge splitting surgery????

DETAILED DESCRIPTION:
PICO P- Horizontal deficient alveolar ridge in Anterior Maxillary Region I- Computer guided surgical cutting guide C- Conventional alveolar ridge splitting O- Clinical outcome and radiographic outcomes Primary outcome: Accuracy In computer Guided: CBCT will performed pre-operative and post-operative for measure the difference of degree in superimposition after ridge splitting.

In conventional method: Ridge mapping will applied in preoperative clinical evaluation, and measure in post-operative, the difference in splitting will calculate in millimeter (mm) Secondary outcome: Thickness of buccal cortical plate In both technique CBCT will performed and measuring the Both Buccal and palatal cortical bone in millimeter(mm)

ELIGIBILITY:
Inclusion Criteria:

* Partial edentulous in the aesthetic zone.
* Patient with bucco-lingual bone width is 3 mm or greater but < 6mm
* Normal alveolar bone height
* Adequate oral hygiene
* Free of soft tissue or dental pathology
* Patients accepting to participate in the study

Exclusion Criteria:

* Patient medically compromised.
* Uncooperative patient.
* Poor oral hygiene and periodontal disease.
* Patients who smoked and pregnant women
* Systemic disease directly affecting bone healing
* Atrophic ridges (1.5 mm or less)
* History of radiotherapy & treatment with bisphosphonates.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy | up to 4 months
  In computer Guided: CBCT will performed pre-operative and post-operative for measure the difference of degree in superimposition after ridge splitting.
  In conventional method: Ridge mapping will applied in preoperative clinical evaluation, and measure in post-operative, the difference in splitting will calculate in millimeter (mm) In computer Guided: CBCT will performed pre-operative and post-operative for measure the difference of degree in superimposition after ridge splitting.
  In conventional method: Ridge mapping will applied in preoperative clinical evaluation, and measure in post-operative, the difference in splitting will calculate in millimeter (mm)

SECONDARY OUTCOMES:
Thickness of buccal cortical plate | up to 4 months
  In both technique CBCT will performed and measuring the Both Buccal and palatal cortical bone in millimeter(mm)

IPD SHARING:
Plan to Share IPD: Undecided